CLINICAL TRIAL: NCT00728572
Title: The Effect of Logan Basic Technique Apex Contact Adjustment on the Motor Recruitment Pattern in the Erector Spinae.
Brief Title: Logan Basic Technique Measured by Surface Electromyography (EMG)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Principal Investigator, Brian Snyder, DC, Research Associate, Logan College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SR0331080126
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Spinal Manipulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Participant will receive a brief exam, a Basic Technique apex contact adjustment and Surface EMG.
  Interventions: Procedure: Logan Basic Technique and Surface EMG; Other: Surface EMG
- Sham (Sham Comparator): Participants will receive a sham Basic Technique adjustment (an adjacent contact not indicated by examination)and surface EMG.
  Interventions: Other: Surface EMG; Procedure: Logan Basic Technique Sham

INTERVENTIONS:
Procedure: Logan Basic Technique and Surface EMG — Participant will receive a brief Basic Technique and Surface EMG examination and Basic Technique treatment.
  Arms: Experimental
Other: Surface EMG — Surface EMG only, no intervention
Procedure: Logan Basic Technique Sham — Participants will receive a sham Basic Technique treatment, not indicated by examination.
  Arms: Sham

SUMMARY:
The purpose of this investigation is to determine the effect of Logan Basic Technique apex contact adjustment (LBT); on the motor recruitment pattern in the erector spinae group via surface EMG.

DETAILED DESCRIPTION:
LBT is a low force adjusting technique that focuses on the foundation segment of the spine, the sacrum, with application of contact on the sacrotuberous ligament which relieves fatigued and strained muscles, particularly intrinsic muscles of the back. Surface electromyography (EMG) is a method of analyzing the activity level of superficial muscles. It is convenient and advantageous when studying muscle relaxation which occurs in biofeedback studies

ELIGIBILITY:
Inclusion Criteria:

* Students in trimesters 1 - 3.
* Naive to the Logan Basic Technique adjusting protocol.

Exclusion Criteria:

* Students in trimesters 4 - 10.
* Pregnant females or females who can possibly be pregnant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Surface EMG | 15 minute sEMG: 5 mins before, 5 mins during and 5 mins after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Logan University, College of Chiropractic, St Louis, Missouri, United States